CLINICAL TRIAL: NCT03771794
Title: Non-Invasive Peripheral Neuromodulation to Augment HRV in Healthy Adults
Brief Title: Heart Rate Variability Augmentation With RR2 Neuromodulation Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Ahud Sternberg, Chairman of Helsinki Ethics Committee, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0024-18-HYMC
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Healthy
Keywords: HRV; Peripheral neuromodulation; Autonomic balance

STUDY DESIGN:
Intervention Model Description: Active Comparator: ReguRate RR2 active. Device: ReguRate neurostimulation system
  Sham Comparator: ReguRate RR2 placebo. Device: Sham ReguRate electrical stimulation - mock sham stimulation mode
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: ReguRate RR2 active (Active Comparator): Device: ReguRate neurostimulation device
  Interventions: Device: ReguRate neurostimulation
- Sham Comparator: ReguRate RR2 sham. (Sham Comparator): Device: Sham ReguRate neurostimulation - mock sham stimulation mode
  Interventions: Device: ReguRate neurostimulation

INTERVENTIONS:
Device: ReguRate neurostimulation — Device: ReguRate neurostimulation Device:
  Sham : ReguRate neurostimulation - mock sham stimulation mode
  Other Names: Sham ReguRate neurostimulation - mock sham stimulation mode

SUMMARY:
Brief Summary: A randomized double-blinded, sham-controlled, crossover study

Condition or Disease: impaired autonomic balance measured by heart rate variability

DETAILED DESCRIPTION:
A randomized double-blinded, sham-controlled, crossover study

Condition or Disease: impaired autonomic balance measured by heart rate variability

Intervention/treatment:

Device: ReguRate RR2 neurostimulation system Device: Sham ReguRate RR2 neurostimulation system

Study Design:

Study Type: Interventional (clinical trial) Planned enrollment: 60 participants Allocation: Randomized Intervention Model; Cross Over Masking: Double (participant, Investigator) Primary Purpose: Treatment Official Title: Non-Invasive peripheral neuromodulation to augment HRV in healthy adults

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion criteria :

1. Healthy male and female volunteers ages 25-60
2. 2 minute HRV measurement with SDNN<35 ms (below 35 ms)
3. Participants able and willing to comply with the study protocol
4. Participants able and willing to sign a written informed consent

Exclusion Criteria:

-

Exclusion criteria :

1. Participant with a known cardiovascular disease
2. Participants with COPD
3. Participants with any known history of epilepsy
4. Participants with detected arrhythmia on test day
5. Participants with implanted electrical and/or neurostimulation device (such as cardiac pace maker/defibrillator/VNS stimulator/SNS stimulator/occipital nerve stimulator/deep brain stimulator etc.)
6. Heavy smokers (more than 1 package of cigarets a day)
7. Participants with a plan to change medications
8. History of vasovagal syncope
9. Pregnancy or bleeding
10. Participants enrolled in another clinical trial

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with 15% or HRV change immediately after neurostimulation session | 1 week
  HRV augmentation

SECONDARY OUTCOMES:
Decrease in heart rate | 1 week
  Percentage of patients with 5% or more decrease in heart rate

OTHER OUTCOMES:
Percentage of patients with 5% or more decrease in blood pressure | 1 week
Percentage of patients with change in additional HRV parameters (rMSSD, LF,HF,L/HF) | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Wingate Institute, Netanya, Israel

IPD SHARING:
Plan to Share IPD: Undecided